CLINICAL TRIAL: NCT06337825
Title: Object Assessment of Improvement in Non-Specific Symptoms After Parathyroidectomy for Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-727
Record Dates: First submitted 2024-03-12; First posted 2024-03-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Primary Hyperparathyroidism; Multinodular Goiter
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 40 patients with primary hyperparathyroidism: patients undergoing parathyroidectomy for primary hyperparathyroidism
  Interventions: Behavioral: Activity Tracker (Fitbit); Diagnostic Test: HbA1C; Behavioral: The PROMPT Questionnaire
- 40 patients with multinodular goiters: patients undergoing thyroidectomy for multinodular goiter
  Interventions: Behavioral: Activity Tracker (Fitbit); Diagnostic Test: HbA1C; Behavioral: The PROMPT Questionnaire

INTERVENTIONS:
Behavioral: Activity Tracker (Fitbit) — Wearable, activity tracker
Diagnostic Test: HbA1C — Average blood glucose (sugar) levels reported as a percentage
Behavioral: The PROMPT Questionnaire — The PROMPT Questionnaire which is a 30-question previously validated assessment for non-specific symptoms in PHPT, will be administered to patients preoperatively and at 2-weeks and 6-months postoperatively

SUMMARY:
Wearable electronic devices are becoming more prevalent in daily life, as they offer real time information on physiological parameters such as heart rate, activity level, oxygenation, and sleep patterns for their users. These wearable electronic devices are easy to install and offer no major risk or discomfort to the user. Implementation of these technologies into medicine has exponentially grown in the past decade with supporting evidence for their use in cardiovascular disease and sleep medicine. The investigators believe that these devices will be able to capture the changes associated with improvement in non-specific symptoms that have not been previously demonstrated.

DETAILED DESCRIPTION:
Primary hyperparathyroidism (PHPT) may be more common than previously assumed.1 Historically, osteoporosis and nephrolithiasis were the only two indications for parathyroidectomy (PTX) based on symptomology.2 All other patients, even in the presence of non-specific symptoms related to PHPT, were not routinely recommended for surgery. Nowadays, however, there is increased understanding that a patient's quality of life (QOL) may be adversely affected by these non-specific symptoms.3 The American Association of Endocrine Surgeons (AAES) strongly recommends PTX in patients with these non-specific symptoms if they can be attributed to PHPT.4 Despite this, these neuropsychiatric, musculoskeletal, and gastrointestinal symptoms are overall difficult to quantify and the improvements in symptoms are mostly measured with QOL surveys.

Even QOL surveys are subjective, and therefore, this may be a major barrier in broadening the indications for parathyroidectomy in patients with PHPT. To this day, there is no proposed objective metrics to quantify these improvements after parathyroidectomy.

Furthermore, the effect of PHPT on cardiovascular risk has been studied, but so far the results are conflicting. The mechanisms for this increased cardiovascular risk are not fully understood.

Nonetheless, this population demonstrates higher rates of hypertension, dyslipidemia, obesity, diabetes, and atherosclerosis compared to the general population. On the other hand, depression and sleep disturbances are also known factors for these comorbidities. It is possible that the neuropsychiatric symptoms of PHPT may contribute to a sedentary lifestyle and thus increase the cardiovascular risk. The association between these two have not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Study group: Consecutive patients older than 18 years old who will undergo PTX for PHPT. The indications and need for surgery will be independent from the research team.
* Control group: Consecutive patients older than 18 years old who will undergo thyroidectomy for multinodular goiter (MNG). The indications and need for surgery will be independent from the research team.

Exclusion Criteria:

* Patients with recurrent or persistent PHPT will not be included.
* Patients who are included but have evidence of recurrent or persistent PHPT based on six-month laboratory workup will be excluded from the final analysis (<5% expected)4.
* Established diagnosis of thyroid cancer or Graves' disease.
* Musculoskeletal or neurologic disorders that affect the patient's activity level.
* Cardiac arrhythmias that would interfere with the wearable electronic device measurement.
* Sleep apnea and other sleep disturbances undergoing concurrent treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred by other physicians for surgical treatment of PHPT and MNG will be identified in the outpatient schedule of our six endocrine surgeons at the Department of Endocrine Surgery, Endocrine and Metabolism Institute. The research team will be introduced to the patients via My Chart where we will request permission for a phone call to discuss the research study. Once they agree to participate, the recruitment will be done at the outpatient clinic in the Endocrine and Metabolism Institute at Main Campus on the day of their appointment. The need for surgery will be made by the treating surgeon with no involvement of the research team. The recruitment will be done by a member of the research team at the endocrine surgery center (F-20).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Change in resting heart rate over time among study participants as monitored by fitness tracker | 7 months
  To assess the change in resting heart rate before and after parathyroidectomy in patients with Primary hyperparathyroidism
Change in number of awakenings during sleep over time among study participants as monitored by fitness tracker | 7 months
  To assess the change in number of awakenings during sleep before and after parathyroidectomy in patients with Primary hyperparathyroidism
Change in % Deep Sleep over Total Sleep Minutes over time among study participants as monitored by fitness tracker | 7 months
  To assess the change in % Deep Sleep over Total Sleep Minutes before and after parathyroidectomy in patients with Primary hyperparathyroidism
Change in steps over time among study participants as monitored by fitness tracker | 7 months
  To assess the change in steps before and after parathyroidectomy in patients with Primary hyperparathyroidism
Change in total active minutes over time among study participants as monitored by fitness tracker | 7 months
  To assess the change in total active minutes before and after parathyroidectomy in patients with Primary hyperparathyroidism
Change in% Active Calorie over Total Calories over time among study participants as monitored by fitness tracker | 7 months
  To assess the change in % Active Calorie over Total Calories before and after parathyroidectomy in patients with Primary hyperparathyroidism
Change in glucose levels (HbA1C) | 7 months
  To assess the change glucose control before and after parathyroidectomy in patients with Primary hyperparathyroidism.
Correlation of Quality of Life surveys with the PROMPT survey | 7 months
  To correlate the measurements of patient health parameters with quality of life surveys before and after parathyroidectomy. This survey is comprised of 30 questions each with a 1 - 5 rating scale where lower scores indicate less pain, fatigue, soreness and higher scores indicate more fatigue, pain, soreness etc.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Jin, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No